CLINICAL TRIAL: NCT02611908
Title: A Phase 1 Clinical Trial to Evaluate Obinutuzumab With High-dose Ibrutinib for the Treatment of Patients With Chronic Lymphocytic Leukemia With Progressive Disease on Single Agent Ibrutinib.
Brief Title: Obinutuzumab With High-dose Ibrutinib for the Treatment of Patients With Chronic Lymphocytic Leukemia With Progressive Disease on Single Agent Ibrutinib.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Michael Choi (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Michael Choi, Assistant Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 151231
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; cancer; obinutuzumab; ibrutinib; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — ibrutinib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ibrutinib +obinutuzumab (Experimental)
  Interventions: Drug: ibrutinib; Drug: obinutuzumab

INTERVENTIONS:
Drug: ibrutinib — Cohort 1 420 mg PO daily Cohort 2 560 mg PO daily Cohort 3 700 mg PO daily Cohort 4 840 mg PO daily
  Other Names: Imbruvica
Drug: obinutuzumab — obinutuzumab 100 mg IV on day 1, 900mg IV on day 2, 1000mg IV day 8, 15, 28 then q 28 days for a total of 8 doses.
  Other Names: Gazyva

SUMMARY:
The purpose of the study is to investigate whether the combination of obinutuzumab and ibrutinib (administered up to 840 mg per day) might be useful for the treatment of CLL or SLL that is not responding or no longer responding to treatment with ibrutinib alone. The study will evaluate whether this regimen can reduce the amount of cancerous cells in the body. Subjects will be treated with ibrutinib at a dose of up to 840 mg a day by mouth, as well as obinutuzumab infusions. Although both of these agents are approved by the FDA for the treatment of CLL or SLL, the combination and the dosing schedule of ibrutinib are considered experimental.

DETAILED DESCRIPTION:
This is phase 1 study for patients with CLL or small lymphocytic lymphoma (SLL) experiencing disease progression on single ibrutinib. This study will evaluate the optimal ibrutinib dose (including doses higher than 420 mg) when combined with obinutuzumab.

During the screening period, patients will continue on ibrutinib at their previous tolerated dose, unless required to stop (e.g.: by a preceding clinical trial).

On cycle 1, day 1, the dose of ibrutinib will be assigned based on the dose cohort. Patients in cohort 1 will receive ibrutinib 420 mg PO daily. Patients in cohort 2 will receive ibrutinib 560 mg PO daily. Cohort 3 will be 700 mg PO daily. Cohort 4 will be 840 mg PO daily.

On cycle 1, day 1, patients will also initiate treatment with obinutuzumab (100 mg on day 1, 900mg on day 2, 1000mg day 8, 15, 28 then q 28 days for a total of 8 doses).

The primary safety endpoint is determination of DLTs during the first 28 days. The primary efficacy endpoint of overall response rate will be assessed 2 months after the final dose of obinutuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and phenotypic verification of B cell CLL or SLL and measurable disease.
* Prior therapy: Patients must have been receiving single agent ibrutinib therapy at the time of disease progression. Patient may have received other therapy in combination with ibrutinib earlier in the their treatment course. Prior obinutuzumab therapy is also permitted.
* Progressive disease on current single agent ibrutinib therapy (but not within the first 2 months of initiating ibrutinib therapy). Progression is based on 2008 iwCLL definition.
* ECOG performance status of 0-2.
* Adequate hematologic function.
* Adequate renal function.
* Adequate hepatic function.

Exclusion Criteria:

* Known CNS lymphoma or leukemia
* History of Richter's or prolymphocytic transformation.
* Primary ibrutinib resistance, defined by progressive disease within the first 2 months of first initiating ibrutinib therapy.
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenia purpura (ITP)
* CLL therapy, with the exception of ibrutinib within the following timeframes:

  1. Chemotherapy, external beam radiation therapy, anticancer antibodies within 30 days prior to the first dose of drug on this study.
  2. Corticosteroid use 20mg prednisone within 1 week prior to first dose on this study.
  3. Radio- or toxin-conjugated antibody therapy within 10 weeks prior to first dose on this study.
  4. Allogeneic stem cell transplant within 6 months prior to first dose on this study
* History of major surgery within 4 weeks prior to first dose on this study.
* History of prior malignancy, with the exception of adequately treated non-melanoma skin cancer, malignancies treated with curative intent and with no evidence of active disease for more than 3 years, or adequately treated cervical carcinoma in situ without current evidence of disease.
* Currently active clinically significant cardiovascular disease or history of myocardial infarction within 6 months of first dose.
* Serologic status and/or PCR testing reflecting active hepatitis B or C infection.
* Known history of infection with human immunodeficiency virus (HIV).
* Unable to swallow capsules or disease significantly affecting gastrointestinal function.
* History of stroke or intracranial hemorrhage within 6 months of first dose.
* Requires anticoagulation with warfarin or other Vitamin K antagonists.
* Requires treatment with a strong CYP 3A inhibitor.
* Pregnant or breast-feeding women
* Women of child-bearing age must obtain a pregnancy test and pregnant or breast feeding females
* Patients who are currently receiving another investigational therapy
* Current infection requiring parenteral antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 2 months

SECONDARY OUTCOMES:
Treatment-emergent adverse events | 2 years
overall response rate | 2 months
progression free survival | 2 months
stable disease rate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — University of California, San Diego